CLINICAL TRIAL: NCT04157153
Title: BIOTRONIK - Safety and Clinical Performance of the - Sirolimus-Eluting Resorbable Coronary Magnesium Scaffold System (DREAMS 3G) in the Treatment of Subjects With de Novo Lesions in Native Coronary Arteries
Brief Title: First in Men Study: BIOMAG-I
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1702
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All subjects will be implanted with the Sirolimus-Eluting Resorbable Coronary Magnesium Scaffold System (DREAMS 3G) and followed up until 60 months.
  Interventions: Device: Implantation of a Sirolimus-Eluting Resorbable Coronary Magnesium Scaffold

INTERVENTIONS:
Device: Implantation of a Sirolimus-Eluting Resorbable Coronary Magnesium Scaffold — Subjects with symptomatic coronary artery disease who qualify for percutaneous coronary intervention (PCI) will be treated with a sirolimus eluting resorbable coronary Magnesium scaffold

SUMMARY:
A prospective, multi-center, first-in-man trial. Up to 115 subjects will be enrolled.

DETAILED DESCRIPTION:
Clinical follow-up visits will take place at 1, 6, and 12 months and annually thereafter until 60 months post procedure.

All subjects will undergo an angiographic follow-up at 6- and 12-month follow up.

IVUS, (including IVUS-VH documentation) and OCT will be performed for all subjects at 6-month and 12-month follow-up (if the safety of the subject allows it and as per the investigator's decision).

Vasomotion will be assessed angiographically with Acetylcholine followed by Nitroglycerine at 12 months follow up in a subgroup of subjects, upon the investigators discretion and if subject consents.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 18 years and < 80 years of age
2. Written subject informed consent available prior to PCI
3. Subject eligible for PCI
4. Subjects with a maximum of two single lesions in two separate coronary arteries which have to be de novo lesions and can be covered with 1 device each
5. Reference vessel diameter between 2.5-4.2 mm by visual estimation, depending on the scaffold size used
6. Target lesion length ≤ 28 mm by visual estimation, depending on the scaffold size used
7. Target lesion stenosis by visual estimation > 50% - < 100% and TIMI flow ≥1 (assisted by e.g. QCA / IVUS /FFR).
8. Subjects with stable or unstable angina pectoris or documented silent ischemia or hemodynamically stable NSTEMI patients without angiographic evidence of thrombus at target lesion
9. Eligible for Dual Anti Platelet Therapy (DAPT)

Exclusion Criteria:

1. Pregnant or breast-feeding females or females who intend to become pregnant during the time of the study
2. Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute ST elevation myocardial infarction (STEMI) within 72 hours prior to the index procedure.
3. Left main coronary artery disease
4. Three-vessels with coronary artery disease requiring treatment at time of procedure
5. Planned interventional treatment of any non-target vessel within 12-month post-procedure
6. Subjects on dialysis
7. Planned intervention of the target vessel post index procedure
8. Ostial target lesion (within 5.0 mm of vessel origin)
9. Target lesion involves a side branch >2.0 mm in diameter
10. Documented left ventricular ejection fraction (LVEF) ≤ 30% within the last 6 months
11. Heavily calcified lesion
12. Target lesion is located in or supplied by an arterial or venous bypass graft
13. Target lesion requiring treatment with a device other than the non-compliant pre-dilatation balloon or scoring balloon prior to scaffold placement (including but not limited to rotational atherectomy, etc.)
14. Unsuccessful pre-dilatation, defined as a residual stenosis rate more than 20%, estimated by any method and/or angiographic complications (e.g. distal embolization, side branch closure, extensive dissections)
15. Known allergies to: Acetylsalicylic Acid (ASA), P2Y12 inhibitors, Heparin, Contrast medium, Sirolimus, or similar drugs; or the scaffold material
16. Subject is receiving an oral or intravenous immuno-suppressive therapy (e.g., inhaled steroids are not excluded) or has a known life-limiting immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus) diabetes mellitus is not excluded)
17. A stenosis located proximal or distal to the target lesion that might require future revascularization or an impede run off detected during diagnostic angiography
18. Life expectancy less than 1 year
19. Planned surgery or dental surgical procedure within 6 months after index procedure unless DAPT will be maintained
20. In the investigators opinion, subject will not be able to comply with the follow-up requirements
21. Subject is currently participating in another study with an investigational device or an investigational drug and has not reached the primary endpoint yet

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
In scaffold late lumen loss | At 6 months after index procedure
  Independent Core Lab Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Haude, Prof, Principal Investigator — Rheinland Klinikum Lukaskrankenhaus Neuss
Locations (14):
- Medizinische Universität Graz, Graz, Austria
- Belgium (3):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - Ziekenhuis Oost-Limburg, Genk
  - UZ Leuven Gasthuisberg, Leuven
- Germany (5):
  - Segeberger Kliniken, Bad Segeberg
  - Herz-und Gefäßzentrum Oberallgäu-Kempten, Kempten
  - Johannes Wesling Klinikum Minden, Minden
  - Deutsches Herzzentrum, Münich
  - Rheinland Klinikum Lukaskrankenhaus Neuss, Neuss
- Onze Lieve Vrouwe Gasthuis Amsterdam (OLVG), Amsterdam, Netherlands
- Miedziowe Centrum Zdrowia SA, Lubin, Poland
- Hospital Clinico San Carlos, Madrid, Spain
- Lund University Hospital, Lund, Sweden
- University Hospital Geneva HUG, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aytekin A, Seguchi M, Xhepa E, Haude M, Wlodarczak A, van der Schaaf RJ, Torzewski J, Garcia-Garcia HM, Waksman R, Joner M. The Impact of Underlying Plaque Characteristics Following the Third-Generation Resorbable Magnesium Scaffold Implantation: An Intravascular OCT Assessment up to 12-Months. Catheter Cardiovasc Interv. 2025 Jun;105(7):1563-1571. doi: 10.1002/ccd.31486. Epub 2025 Mar 16. PMID 40091374
- [Derived] Haude M, Wlodarczak A, van der Schaaf RJ, Torzewski J, Ferdinande B, Escaned J, Iglesias JF, Bennett J, Toth GG, Joner M, Toelg R, Wiemer M, Olivecrano G, Vermeersch P, Garcia-Garcia HM, Waksman R. A new resorbable magnesium scaffold for de novo coronary lesions (DREAMS 3): one-year results of the BIOMAG-I first-in-human study. EuroIntervention. 2023 Aug 7;19(5):e414-e422. doi: 10.4244/EIJ-D-23-00326. PMID 37334655
- [Derived] Haude M, Wlodarczak A, van der Schaaf RJ, Torzewski J, Ferdinande B, Escaned J, Iglesias JF, Bennett J, Toth G, Joner M, Toelg R, Wiemer M, Olivecrona G, Vermeersch P, Garcia-Garcia HM, Waksman R. Safety and performance of the third-generation drug-eluting resorbable coronary magnesium scaffold system in the treatment of subjects with de novo coronary artery lesions: 6-month results of the prospective, multicenter BIOMAG-I first-in-human study. EClinicalMedicine. 2023 Apr 17;59:101940. doi: 10.1016/j.eclinm.2023.101940. eCollection 2023 May. PMID 37113674